CLINICAL TRIAL: NCT05580978
Title: Libre 2 CGM Plus Glycemic Excursion mIniMization (GEM) in the Treatment of PrEDiabEtes
Brief Title: CGM Plus GEM in Prediabetes
Acronym: IMPEDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Abbott Diabetes Care (Industry); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 21-4931
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: PreDiabetes
Keywords: prediabetes; lifestyle guide; continuous glucose monitor; prevention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GEM + CGM + Activity Monitor (Experimental): GEM plus CGM and Activity Monitor (FitBit)
  Interventions: Behavioral: GEM
- Routine Care (Active Comparator): Usual care already being received for prediabetes as treated by their care team.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: GEM — The intervention group will be given Libre 2 supplies for 4 months, an activity monitor, and the 4-chapter GEM paper guide. The intervention group will complete a virtual or inperson study visit where they will receive instructions on how to apply their unblinded Freestyle Libre and connect it to the study account, as well as how to register their Fitbit to the study account. Participants will receive one telephone call to review use of the GEM Guide and call at two weeks and six weeks later when the probability of dropouts from lifestyle intervention peaks. Participants will follow the self-directed GEM guide for 4 months (a 1-month treatment period followed by a 3-month maintenance period) while wearing a FitBit activity monitor and a Freestyle Libre 2 CGM.
  Arms: GEM + CGM + Activity Monitor
Other: Routine Care — Participant's current prediabetes treatment.
  Arms: Routine Care

SUMMARY:
This study is designed to look into the effect of a lifestyle management guide called GEM (Glycemic Excursion Minimization) alongside continuous glucose monitoring (CGM) and an activity monitor (FitBit) and the effect this can have on persons with prediabetes.

DETAILED DESCRIPTION:
For people with prediabetes, it may be possible to delay or prevent the progression to diabetes by reducing postprandial glucose (PPG). The Glycemic Excursion Minimization (GEM) lifestyle intervention guide can reduce PPG in people with type 2 diabetes and has been studied in this population with continuous glucose monitor (CGM) feedback to help the user learn what elevates and lowers their PPG. This study examines if the GEM lifestyle intervention guide plus continuous feedback from the FreeStyle Libre 2 CGM and FitBit will allow participants with prediabetes with HbA1c 6.0-6.4% to (1) improve their metabolic status by illustrating the effects of their routine food and physical activity choices on their glucose levels and variability, more than Routine Care (RC), and (2) to enhance these investigations by adding comprehensive plasma proteomics to the analyses. The investigators will recruit up to 36 adult participants with prediabetes through the University of Colorado, with the goal of having at least 30 participants complete the study. Participants will be randomized to the intervention or RC. Those randomized to the intervention will be given a GEM treatment manual, Libre2 CGM, and an activity monitor and will follow the GEM lifestyle intervention guide for 4 months. Those participants randomized to RC will follow recommendations from their primary care provider. RC participants will have the opportunity to receive GEM four months after consenting and completing the RC pre-post assessments if they meet eligibility criteria. It is anticipated that 50% of the RC participants will want/be able to cross over to GEM upon completion of RC. Pre-post blinded CGM data and activity data, clinical, and psychosocial outcomes will be collected and analyzed. It is anticipated that this pilot project will demonstrate the benefits of using GEM plus FreeStyle Libre 2 and FitBit to reduce percentage of CGM readings >120 mg/dL, from blinded pre-post FreeStyle Libre Pro, as well as reduce BMI and depressive symptoms and increase modified diabetes empowerment. Comprehensive proteomics will be measured on small samples of EDTA treated venous blood. Individual proteins and protein pathways will be measured for each of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-70 years
* A1C 6.0-6.4
* Documented diagnosis of prediabetes
* Have a smart phone
* Able to read English, as the GEM guide is currently only available in English
* Willing and able to follow the study procedures as instructed

Exclusion Criteria:

* Diagnosis of diabetes mellitus
* Currently taking any diabetes medication
* Currently taking medication that promotes insulin resistance or otherwise interferes with metabolic control (e.g., prednisone)
* Has a condition that precludes a low carbohydrate diet, such as gastroparesis
* Has a physical or medical condition that precludes walking 120 steps per minute for 10 minutes or longer
* Has documented kidney disease that would preclude participation in study per PI discretion
* Active or planned cancer treatment
* Extreme visual or hearing impairment that would impair ability to use real-time CGM
* Pregnant or anticipates becoming pregnant in the next 4 months
* Anticipates moving within the next 4 months
* Treating physician, for any reason, considers their patient inappropriate for the study (e.g., uncontrolled bipolar disease)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in percentage of CGM glucose readings > 120 mg/dL | 4.5 months
  Change in percentage of CGM glucose readings > 120 mg/dL from pre-intervention blinded CGM to post-intervention blinded CGM.

SECONDARY OUTCOMES:
Change in HbA1c | 4.5 months
  Change in HbA1c from baseline to post-intervention.
Change in Glucose Variability | 4.5 months
  Change in glucose variability (GV%) as measured by CGM, from baseline to post-intervention.
Change in Body Mass Index | 4.5 months
  Change in Body Mass Index (BMI) from baseline to post-intervention.
Change in Cardiovascular Risk | 4.5 months
  Change in cardiovascular risk as calculated by a validated risk calculator from baseline to post-intervention
Change in Empowerment | 4.5 months
  Change in empowerment as measured by modified Diabetes Empowerment Scale, from baseline to post-intervention.
Change in Depressive Symptoms | 4.5 months
  Change in depression score as measured by PHQ-8 at baseline and post-intervention.
Change in Diabetes Knowledge | 4.5 months
  Change in diabetes knowledge as measured by a modified Diabetes Knowledge Scale from baseline to post-intervention.
Dietary Habits | 4.5 months
  Change in dietary habits as measured by Carbohydrate Routine Consumption Scale from baseline to post-intervention.
Motivation and Attitudes Toward Changing Health | 4.5 months
  Change in Motivation and Attitudes Toward Changing Health (MATCH) score from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Oser, MD, Principal Investigator — Associate Professor, Dept. Family Medicine
Locations (1):
- University of Colorado- Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No